CLINICAL TRIAL: NCT06361160
Title: Reduction of Auditory-Verbal Hallucinations in Schizophrenia Through Cortical Neuromodulation: Towards a Closed-loop System
Brief Title: Reduction of Auditory-Verbal Hallucinations in Schizophrenia Through Cortical Neuromodulation
Acronym: HALLUSTIM
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Centre Hospitalier St Anne (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: Triple | Purpose: Treatment
Other Study IDs: D23-P037
Record Dates: First submitted 2024-03-29; First posted 2024-04-11 (Actual); Last update posted 2024-07-29 (Actual); Status verified 2024-07

CONDITIONS: Treatment Resistant Schizophrenia
Keywords: Treatment Resistant Schizophrenia; Transcranial Magnetic Stimulation (TMS)
MeSH Terms: conditions — Schizophrenia, Treatment-Resistant

STUDY DESIGN:
Intervention Model Description: Patients (20) suffering from resistant schizophrenia will be enrolled over a 12-month period and will be randomized in a (1:1) ratio to start with either active or sham Transcranial Magnetic Stimulation (TMS) for the first of their 12 sessions, which will then alternate from one condition to the other for each patient.
Who Masked: Participant, Care Provider, Outcomes Assessor
Masking Description: Only the person conducting the experiment will know which condition each patient is in.
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Active TMS sessions (Active Comparator): For a given patient, the 6 sessions (out of 12) in which the TMS is active.
  Interventions: Device: Active Transcranial Magnetic Stimulation (TMS)
- Sham TMS sessions (Sham Comparator): For a given patient, the 6 sessions (out of 12) in which the TMS is a sham.
  Interventions: Device: Sham Transcranial Magnetic Stimulation (TMS)

INTERVENTIONS:
Device: Active Transcranial Magnetic Stimulation (TMS) — Active rTMS (continuous theta burst, cTBS) applied to the temporo-parietal junction (TPJ) at the onset of the Auditory Verbal Hallucinations (AVH).
  Other Names: Active TMS
  Arms: Active TMS sessions
Device: Sham Transcranial Magnetic Stimulation (TMS) — Sham rTMS (continuous theta burst, cTBS) applied to the temporo-parietal junction (TPJ) during the onset of the Auditory Verbal Hallucinations (AVH).
  An electrical stimulator is synchronised with the magnetic stimulation to recreate the tactile sensation and the coils emits the same noise during sham stimulation as in the active configuration, making it impossible to distinguish between active and placebo magnetic stimulation.
  Other Names: Sham TMS
  Arms: Sham TMS sessions

SUMMARY:
Approximately 1% of the general population will be affected by schizophrenia over the course of their lives, with life expectancy being reduced by 20 years on average and quality of life being severely diminished in affected individuals. One third of patients suffering from schizophrenia will evolve towards a resistant form of the disease, amongst which many will suffer from auditory-verbal hallucinations (AVH) that current therapeutic approaches struggle to alleviate. Previous work from our team has demonstrated the possibility of robustly inferring the periods of occurrence of AVH from fMRI data, paving the way for the development of a closed-loop neuromodulation system comprised of an electrode array positioned in Broca's area, which would detect AVH in real time, and effector electrodes which would stimulate the temporo-parietal cortex to interrupt them. The aim of this project is to assess the feasibility of this system. To do so, we will first test the ability of transcranial magnetic stimulation of the "continuous theta burst" (cTBS) type, applied at the time of AVH onset, to reduce their duration and intensity, and assess whether this is associated with therapeutic response to the current gold standard rTMS protocol for AVH reduction through neuroplasticity induction. Demonstrating the feasibility of acute suppression of AVH by cortical neurostimulation is an essential element in the feasibility of a closed-loop reactive neuromodulation system.

The research project comprises two phases:

-Phase 1: randomized controlled clinical trial (1 weekly session per patient over 12 weeks: 6 active stimulation sessions and 6 sham sessions) evaluating the phasic effects of rTMS on AVHs as they appear during the sessions.

Phase 2: open-label study offering patients a routine rTMS protocol which has demonstrated its effects on AVH (10 TMS sessions over one workweek - twice daily with 1-hour intervals, MULTIMODHAL study, NCT01373866).

ELIGIBILITY:
Inclusion Criteria:

* Age > 18 years old
* Schizophrenic Disorder (Diagnostic and statistical manual of mental disorders, DSM-5-TR, American Psychiatric Association, 2013)
* AVHs that have resisted to at least two properly conducted antipsychotic therapies at an effective dose for at least 8 weeks (criteria of Kinon et al., 1993)
* Frequent AVHs (at least 10 times per hour) (Fovet et al., 2022)
* Unmodified antipsychotic dosage for 30 days prior to inclusion in the protocol
* AVH are the main residual symptom of schizophrenia.
* Consent to participate in the study

Exclusion Criteria:

* Pregnancy (based on date of last menstrual period with possibility of urine test if in doubt)
* Anticonvulsant therapy
* Neurological disorder (e.g., multiple sclerosis, epilepsy)
* Current addictive behavior (except tobacco and cannabis, widely used in this clinical population; Fovet et al., 2022)
* Contraindication to MRI (i.e., presence of ferromagnetic material or implanted neurostimulation devices due to the risk of displacement or dysfunction such as cochlear implants, cardiac pacemakers, metal splinters in the body following an accident, permanent makeup applied less than 6 months ago, neurosurgical clips, deep brain or vagus nerve stimulation devices, baclofen pumps) (Lefaucheur et al., 2011)
* Morphological criteria: weight > 130 Kg, abdominal circumference conditioned by the opening of the magnet, shoulder width
* Lack of coverage by the social security system
* Current participation in another interventional research protocol or being in the exclusion period of a previous research protocol
* Refusal to be informed of an brain anomaly detected in the MRI
* Person under guardianship or curatorship
* Behavioral disorders or delusions likely to prevent the MRI or rTMS from being performed under good conditions (left to the discretion of the investigator at baseline).

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 20 (Estimated)
Dates: Start 2024-05-21 (Actual); Primary Completion 2026-05 (Estimated); Study Completion 2026-05 (Estimated)

PRIMARY OUTCOMES:
Duration of auditory-verbal hallucinations | During the intervention of Phase 1 (for each active or sham TMS session)
  The primary endpoint is the reduction in the duration of AVH (in seconds) during active phasic stimulation sessions compared to sham sessions. Participants will press a button when an AVH occurs (starting the intervention) and press another when the AVH disappears. This allows for the recording of the duration of the AVHs.

SECONDARY OUTCOMES:
Clinical scales scores | At baseline (before Phase 1), before the intervention of Phase 2 (Day 0, two weeks after the end of Phase 1), after the intervention of Phase 2 (Day 15, Month 1, Month 3, Month 6, Month 12)
  An evaluation of the following clinical measures will take place : AHRS, CGI, Visual analog scale for AVH intensity and frequency, GAF and PANSS.
Measure of the duration and/or intensity of HAV (in seconds) during active phasic stimulation sessions compared to sham sessions (phase 1) among TMS responders and non-responders in phase 2 | Through study completion, an average of 2 years
  Reduction in duration and/or intensity of HAV (in seconds) during active phasic stimulation sessions compared to sham sessions (phase 1) among TMS responders and non-responders in phase 2 (response: decrease in pre/post AHRS score >25%).
Intensity of auditory-verbal hallucinations | During the intervention of Phase 1 (for each active or sham TMS session)
  Phase 1 At the end of each active or sham cTBS train, the computer screen will display an 5-point Likert Scale, through which the patient will have to report AVH-intensity before the session can continue.

CONTACTS AND LOCATIONS:
Overall Officials: Philippe Domenech, MD, PhD, Principal Investigator — GHU Paris Psychiatry & Neurosciences
Locations (1):
- Groupe Hospitalo-Universitaire Paris Psychiatrie & Neurosciences, Paris, France